CLINICAL TRIAL: NCT04352244
Title: The Physiology of Human Brown Adipose Tissue
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Joslin Diabetes Center (Other); Chan Zuckerberg Initiative (Other)
Responsible Party: Principal Investigator, Mary Elizabeth Patti, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2009P-000101
Record Dates: First submitted 2020-03-31; First posted 2020-04-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Adipose Tissue, Brown; Adipose Tissue; Obesity
Keywords: Human Cell Atlas
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Specimens to be retained: blood and adipose tissue samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Participants: Individuals undergoing abdominal surgery or radiologically-guided biopsies for clinical indications will be recruited prior to the planned procedures.
  Interventions: Procedure: Fat biopsy; Diagnostic Test: Blood sampling; Genetic: Blood sample for DNA analysis

INTERVENTIONS:
Procedure: Fat biopsy — The fat biopsy is performed during a scheduled procedure at the Beth Israel Deaconess Medical Center (BIDMC). Routine preoperative procedures will be followed, including local anesthesia (numbing a particular region of the body) or general anesthesia (being put to sleep).
  Adipose tissue will be sampled from different depots depending on the procedure. For example, the surgeon will collect adipose tissue from the neck and supraclavicular depots from cervical spine, thyroid, and parathyroid procedures; perinephric fat from adrenalectomies, omental fat from abdominal procedures, and paraspinal fat from lumbar spine procedures. Up to 5 pieces of fat tissue weighing about three to six grams will be removed. All other aspects of the surgical procedure will proceed as planned. Samples will be prepared for subsequent laboratory analysis.
Diagnostic Test: Blood sampling — A blood sample will be collected in the fasting state either during preoperative testing or in the preoperative area on the day of planned procedure for measurement of adipose functional markers (leptin, adiponectin) and insulin resistance (insulin, C-peptide), and measures of glycemia (glucose, hemoglobin A1c).
Genetic: Blood sample for DNA analysis — Targeted resequencing of DNA to identify variants associated with adipose phenotypes will be performed.

SUMMARY:
Brown fat is a type of fat, found in both children and adults, which can produce heat and regulate the body's metabolism and energy use. White fat is the more common type of fat which is used to store extra calories. Understanding more about differences between brown and white fat may allow us to develop new approaches to improve the body's metabolism.

DETAILED DESCRIPTION:
The overarching goal of this study, is to map fat (adipose) tissue differences in humans. The investigators will probe multiple aspects of fat cell (adipocyte) identity by integrating quantitative chemical imaging, single-cell and single-nucleus RNA sequencing (sc and snRNAseq), and site-specific collection of adipocytes and adipocyte precursors.

Deidentified data from these studies will be submitted to the Human Cell Atlas. The investigators anticipate that these studies will ultimately increase understanding of mechanisms by which fat (adipose) tissue regulates systemic metabolism (energy transformation in the body), and promotes risk for metabolic disease. Knowledge gained from this research may be used to set the stage for disease-specific analyses, and aid in the development of personalized medicine for metabolic diseases such as type 2 diabetes.

ELIGIBILITY:
Inclusion criteria:

1. Healthy participants between age 18 and 75 years undergoing planned clinically indicated procedure at BIDMC.

Exclusion Criteria:

1. Body mass index (BMI) greater than or equal to 40 kg/m2
2. History of any local or systemic infectious disease with fever or requiring antibiotic within four weeks of drug administration;
3. Diabetes, either previously diagnosed or hemoglobin A1c greater than or equal to 6.5%
4. Use of oral or parenteral corticosteroids (epidural permitted) or other medication known to cause insulin resistance in the previous 6 weeks.
5. Willingness to provide informed consent and follow study procedures, including attending scheduled visits.
6. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
7. Hepatic disease, including serum alanine aminotransferase (ALT) or aspartate transaminase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
8. Active malignancy (except squamous or basal cell carcinoma of skin)
9. Bleeding disorder, treatment with anticoagulants (if not discontinued prior to surgery), or platelet count <50,000;
10. Current addiction to alcohol or substances of abuse;
11. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation;
12. Use of an investigational drug within 30 days prior to screening.
13. There will be no involvement of special vulnerable populations such as fetuses, neonates, pregnant women, children, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.
14. Because the goal is to study adult human brown adipose tissue, children are not eligible to participate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants planning a procedure will be recruited from clinical practices of Dr. Andrew White, Dr. Peter Mowschenson, and Dr. Per-Olof Hasselgren at BIDMC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Collect human brown and white adipose tissue to prepare progenitor and differentiated cells for single nucleus RNA analysis. | March 2022
  Adipose tissue biopsy samples will be processed for single-nucleus RNA analysis of gene expression.
Collect human brown and white adipose tissue to prepare progenitor and differentiated cells for Raman spectroscopy. | March 2022
  Adipose tissue biopsy samples will be processed for Raman spectroscopy analysis.
Collect human brown and white adipose tissue to prepare cells for ex vivo differentiation | March 2022
  Adipose tissue biopsy samples will be processed for ex vivo differentiation.
Insulin resistance | March 2022
  Insulin resistance of participants, assessed by homeostatic model of insulin resistance (HOMA-IR), will be analyzed and summarized.
Hemoglobin A1c | March 2022
  Hemoglobin A1c levels for participants will be analyzed and summarized.
Fasting glucose levels | March 2022
  Fasting glucose levels for participants will be analyzed and summarized.
Body mass index (BMI) | March 2022
  Weight and height will be combined to report BMI in kg/m^2. BMI of participants will be analyzed and summarized.
Demographic characteristics | March 2022
  Demographic characteristics of participants will be analyzed and summarized.

SECONDARY OUTCOMES:
DNA analysis | March 2022
  DNA will be isolated and stored from blood samples. If specific genes are differentially regulated as a function of metabolic state or anatomical location of biopsy, locus-specific or genome-wide genotyping may be performed to assess potential regulatory single-nucleotide polymorphisms (SNP).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared with other researchers with permission of local institutional review boards via the Human Cell Atlas database.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of study results
Access Criteria: Data will be shared with academic investigators with approval of local institutional review boards.

DOCUMENTS (1):
  • Informed Consent Form (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT04352244/ICF_000.pdf